CLINICAL TRIAL: NCT04379934
Title: Functional and Metabolic Effects of Ketone Bodies on Human Atrial Tissue in Patients With and Without Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KetoCard01
Record Dates: First submitted 2020-04-30; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure; Ischemia Reperfusion Injury; Mitochondrial Pathology
MeSH Terms: conditions — Heart Failure; Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart failure (Other): Ejection fraction < 45%
  Interventions: Dietary Supplement: 3-hydroxybuturate
- Non-heart failure (Other): Ejection fraction > 45%
  Interventions: Dietary Supplement: 3-hydroxybuturate

INTERVENTIONS:
Dietary Supplement: 3-hydroxybuturate — 3-hydroxybuturate will be administered directly as a modified Krebs Henseleit buffer in a super perfused atrial strips model

SUMMARY:
This proof of concept study aims to evaluate the effects of applying ketone bodies to human atrial tissue biopsies using an atrial strips model and high resolution respirometry.

DETAILED DESCRIPTION:
Ketone bodies are high energy molecules which are naturally occurring in the body during fasting or stress.

Recently, ketone bodies have been shown to improve cardiac function in patients with heart failure(1) through a mechanism, which has yet to be elaborated.

We wish to evaluate the effects of ketone body administration on cardiac tissue subjected to ischemia reperfusion injury. We will evaluate contractile force of the and the mitochondrial performance. Cardiac atrial tissue will be obtained from patients undergoing coronary artery bypass grafting (CABG) or valve replacement surgery. Patients will be recruited after signing an informed consent and allocated in heart failure / non-heart failure groups based on a clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* EF < / > 45%, hospitalized for elective CABG or heart valve surgery

Exclusion Criteria:

* Myocardial infarction within 4 weeks, atrial fibrillation, medically treated thyroid disease, oral treatment with opioids.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Contractile force recovery | Outcome will be assessed within a year when the inclusion of patients is complete
  Atrial strips model, contractile force (nm*mm^-1) during stabilization, ischemia and reperfusion

SECONDARY OUTCOMES:
Mitochondrial respiratory capacity | Outcome will be assessed within a year when the inclusion of patients is complete
  High Resolution Respirometry, Complex I and Complex I+II respiration (pmol O2 · s-1·mg-1) assessed via a substrate and inhibitor (SUIT) protocol.
Mitochondrial Reactive Oxygen Species production | Outcome will be assessed within a year when the inclusion of patients is complete
  High Resolution FluoRespirometry, Complex I and Complex I+II linked ROS generation measured with AmplexUltra red and H2O2 interaction fluorescense

CONTACTS AND LOCATIONS:
Overall Officials: Hans Erik Bøtker, M.D., Prof., Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nielsen R, Moller N, Gormsen LC, Tolbod LP, Hansson NH, Sorensen J, Harms HJ, Frokiaer J, Eiskjaer H, Jespersen NR, Mellemkjaer S, Lassen TR, Pryds K, Botker HE, Wiggers H. Cardiovascular Effects of Treatment With the Ketone Body 3-Hydroxybutyrate in Chronic Heart Failure Patients. Circulation. 2019 Apr 30;139(18):2129-2141. doi: 10.1161/CIRCULATIONAHA.118.036459. PMID 30884964